CLINICAL TRIAL: NCT04424602
Title: Comparison Between Mycophenolate andCyclophosphamide in the Treatment of Lupus Nephritis
Brief Title: Comparison between2 Drugs in Lupus Nephritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, suzan.D.zakaria, principal investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0000085
Record Dates: First submitted 2020-05-02; First posted 2020-06-11 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — Mycophenolic Acid

STUDY DESIGN:
Intervention Model Description: This study will be carried on40 patients with systemic lupus erythematous with lupus nephritis.the age group of patients will be between 20 to50 years.All lupus nephritis patients will be divided randomly into two groups. First group will be 20female patients on lupus nephritis .They will be given oral corticosteroid( 1mg/kg per day) and intra venous cyclophosphamide 500mg once every two weeks for 6months. Second group will be 20female patients on lupus nephritis they will be given oral corticosteroid(1mg/kg per day) and oral mycophenolat 2 to 3mg/kg for 6 months
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cyclophosphamide (Experimental): participants will receive intra venous cyclophosphamide 500mg once every two weeks for 6months.
  Interventions: Drug: cyclo phosphamide
- mycophenolate (Active Comparator): participants will receive oral mycophenolat 2 to 3mg/kg for 6 months.
  Interventions: Drug: mycophenolate

INTERVENTIONS:
Drug: cyclo phosphamide — 500mg vial
  Arms: cyclophosphamide
Drug: mycophenolate — 500mg film-coated tablets.
  Arms: mycophenolate

SUMMARY:
The aim of this work is to study the effect and side effects of the cyclophosphamide versus mycophenolate in lupus nephritis

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE), also known simply as lupus, is an autoimmune disease in which the body's immune system mistakenly attacks healthy tissue in many parts of the body.

Symptoms vary between people and may be mild to severe. common symptoms include painful and swollen joints, fever, chest pain, hair loss, mouth ulcers, swollen lymph nodes, feeling tired, and a red rash which is most commonly on the face. Often there are periods of illness, called flares, and periods of remission during which there are few symptoms.painless passage of blood or protein in the urine may often be the only presenting sign of kidney involvement.

Acute or chronic renal impairment may develop with lupus nephritis, leading to acute or end-stage kidney failure. Because of early recognition and management of SLE, end-stage renal failure occurs in less than 5% of cases; except in the black population, where the risk is many times.Nephritis is the most severe manifestation of lupus. Between 1950s and 1970s, corticosteroids were used for the treatment of lupus nephritis (LN) ,and using of cyclophosphamide(CPM), improved the outcome dramatically with 5 years survival increasing from 17% to 80%.Subsequently, intravenous (iv) CPM became the standard of care in induction regimes; however, ivCPM was associated with complications such as bladder toxicity, gonadal problems, and infections. To reduce the toxicity, low-dose of 500mg iv(CPM) every two weeks for six months showed equivalent efficacy and less side effect.

Mycophenolatemofetil(MMF) is widely used in solid organ transplantation and it reduces the rate of acute rejection following renal transplantation.

It has also been used to treat patients with other immune-mediated disorders such as immunoglobulin A nephropathy, small-vessel vasculitides and psoriasis .

Lupus nephritisis inflammation of the kidney that is caused by systemic lupus erythematous (SLE). Lupus nephritis happens when lupus involves the kidneys.its symptoms, though, are not always dramatic. for many, the first noticeable symptom is swelling of the legs, ankles and feet. less often, there can be swelling in the face or hands.

ELIGIBILITY:
Inclusion Criteria:

1. All patients have systemic lupus erythromatosis with lupus nephritis either newly diagnosed or with history of SLE with lupus nephrits
2. All stage of lupus nephritis except stage(i,v,vi)
3. patients who accepted to participate in the study.

Exclusion Criteria:

1. Patient with acute inflammatory process such as(rheumatoid arthritis or other rhumatoligical diseases).
2. Patients who are taking other immunosuppressive therapy.
3. Patients with malignancies.
4. Patients with HCV, HBV or HIV infection.
5. Patients with lupus nephritis sage(i,v,vi).

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2021-09-05 (Actual); Study Completion 2021-09-09 (Actual)

PRIMARY OUTCOMES:
serume creatinine (sCR) | 6 months
  to measure treatment response and determine renal function These investigation will be done before starting the pharmacotherapy and after the end of the therapy.its normal range from(0.4 to1.5 mg/dl)its level increase in lupus.
blood uerea nitrogen. | 6 months
  to measure treatment response and determine renal function These investigation will be done before starting the pharmacotherapy and after the end of the therapy.its normal range ,around7to20mg/dl(2.5to7.1mmol) its level increase in lupus.
• Erythrocyte sedimentation rate.(ESR) | 6 months.
  can help us to determine if patients have inflammation.These investigation will be done before starting the pharmacotherapy and after the end of the therapy .its range from (15to10mm/hr)its level increase in lupus.
• Anti ds DNA | 6 months
  will done for diagnosis and ascertain activity of lupusThese investigation will be done before starting the pharmacotherapy and after the end of the therapy if the antidsDNA level are high the lupus may be active and if its level is low the lupus is less active.its rangr(<18iu/ml)
• Complement 3 (C3) | 6 months
  will done for diagnosis and ascertain activity of lupus These investigation will be done before starting the pharmacotherapy and after the end of the therapy .c3range from75to175mg/lcomplementc3 level are lower in lupus.
• complete blood count.(CBC)( red blood cells,white blood cells,platelets) | 6 months
  to know all information about red blood cells,white blood cells,platelets and effect of two drus on it.These investigation will be done before starting the pharmacotherapy and after the end of the therapy at six months.
• 24h urine test for creatinine clearance and protien excretion. | 6 months.
  the test is used to check kideny function.•These investigation will be done before starting the pharmacotherapy and after the end of the therapy.normal urinary protie-to-creatinine ratio is<0.2.

CONTACTS AND LOCATIONS:
Locations (1):
- ALAzhar university, Cairo, Egypt